CLINICAL TRIAL: NCT00668109
Title: A Randomized, Open-label, Multi-center, Parallel Group Study to Investigate the Efficacy and Safety of Vardenafil in Comparison to Tadalafil in Males With Erectile Dysfunction and a Diagnosis of Diabetes, Hypertension or Hyperlipidemia
Brief Title: Assessment of Efficacy of Vardenafil in Subjects With Erectile Dysfunction and Diabetes, Hypertension or Hyperlipidemia
Acronym: LUTECIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10893
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Diabetes mellitus; Hypertension; Hyperlipidemia; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus; Hypertension; Hyperlipidemias | interventions — Vardenafil Dihydrochloride; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Active Comparator)
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 10 mg one hour prior to sexual intercourse
  Arms: Arm 1
Drug: Tadalafil — 10 mg taken approximately 24 hours prior to sexual intercourse
  Arms: Arm 2

SUMMARY:
Assessment of efficacy of vardenafil in subjects with erectile dysfunction and diabetes, hypertension or hyperlipidemia

ELIGIBILITY:
Inclusion Criteria:- Age: 18 years and older- Males with erectile dysfunction- Stable heterosexual relationship- Medical history / diagnosis of diabetes mellitus and/or hypertension and/or hyperlipidemia Exclusion Criteria:- Primary hypoactive sexual desire- History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months- Nitrate use- Other exclusion criteria apply according to Summary of Product Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2003-12; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Sexual encounter profile question 3 observed within 15 minutes to 4 hours for vardenafil and 22 to 26 hours for the tadalafil group | 4 weeks

SECONDARY OUTCOMES:
Sexual encounter profile question 2 | 4 weeks
Hardness of erection | 4 weeks
Other diary based variables | 4 weeks
Safety and tolerability | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (62):
- Belgium (3):
  - Bruxelles - Brussel
  - Edegem
  - Roeselare
- Colombia (4):
  - Barranquilla
  - Bogotá
  - Medellín
  - Santa Fé de Bogotá
- Finland (2):
  - Helsinki
  - Oulu
- Germany (12):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Stuttgart, Baden-Wurttemberg
  - Königsbrunn, Bavaria
  - München, Bavaria
  - Weiden, Bavaria
  - Hamburg, Hamburg
  - Marburg, Hesse
  - Hanover, Lower Saxony
  - Osnabrück, Lower Saxony
  - Westerstede, Lower Saxony
  - Mönchengladbach, North Rhine-Westphalia
  - Berlin, State of Berlin
- Israel (4):
  - Haifa, Israel
  - Jerusalem, Israel
  - Tel Aviv, Israel
  - Tel Litwinsky
- Italy (6):
  - Catania
  - Milan
  - Padua
  - Pavia
  - Perugia
  - Pisa
- Mexico (5):
  - Durango, Durango
  - Iguala de la Independencia, Guerrero
  - México, D. F., México, D. F.
  - Monterrey, Nuevo León
  - México, D.F.
- Netherlands (2):
  - Nijverdal
  - Utrecht
- Norway (4):
  - Moelv
  - Oslo
  - Sarpsborg
  - Trondheim
- Peru (2):
  - Callao
  - Lima
- South Africa (7):
  - George, Eastern Cape
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Newcastle, KwaZulu-Natal
  - Pietermaritzburg, KwaZulu-Natal
  - Cape Town, Western Cape
- Spain (8):
  - A Coruña, A Coruña
  - Sant Joan d'Alacant, Alicante
  - L'Hospitalet de Llobregat, Barcelona
  - Castellon, Castellón de La Plana
  - Málaga, Málaga
  - Palma de Mallorca, Palma de Mallorca
  - Vigo, Pontevedra
  - Zaragoza, Zaragoza
- Sweden (3):
  - Borås
  - Skövde
  - Stockholm